CLINICAL TRIAL: NCT06362408
Title: Effect of Intraoperative Use of Dexmedetomidine on Postoperative Mental Disorders and Long-term Survival in Elderly Patients Undergoing Non-cardiac Surgery
Brief Title: Effect of Dexmedetomidine on Postoperative Mental Disorders and Long-term Survival in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fudan University (Other); Peking University People's Hospital (Other); The First Xiangya Hospital of Central South University (Unknown); Second Xiangya Hospital of Central South University (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-DEX-PSM/IPTW-001
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Cohort Studies
Keywords: Dexmedetomidine; Postoperative mental disorders; Long-term survival; Elderly patients; depression; anxiety; delirium
MeSH Terms: conditions — Depression; Anxiety Disorders; Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the DEX group: used DEX (safe use range: 0.2~1.0 μg/(kg·h)) for anesthesia induction or maintenance during surgery
  Interventions: Drug: Dexmedetomidine
- the Non-DEX group: did not use DEX throughout the entire anesthesia process

INTERVENTIONS:
Drug: Dexmedetomidine — Older patients who have used dexmedetomidine(safe use range: 0.2~1.0 μg/(kg·h)) for anesthesia induction or maintenance during surgery were classified as the DEX group. On the contrary, patients who did not use dexmedetomidine throughout the entire anesthesia process were identified as the Non-DEX group.
  Groups: the DEX group

SUMMARY:
China's aging population is causing an increase in the number of senior persons undergoing surgery. More and more clinicians are paying attention to the postoperative survival and mental health of elderly surgical patients.

Dexmedetomidine (DEX) is an alpha-2 adrenergic agonist that works by inhibiting norepinephrine releasing renaline, which reduces inflammation and thus plays a protective role in the central nervous system. DEX has the potential to prevent and treat postoperative anxiety and depression in elderly patients undergoing non-cardiac surgery.

Further exploration of evidence for evidence-based medicine is needed. Based on the above research background, this hypothesis is proposed: in elderly patients undergoing noncardiac surgery, intraoperative DEX is associated with a reduction in short-term postoperative mental disorders and a reduction in long-term postoperative mortality.

DETAILED DESCRIPTION:
Studies have suggested that continuous infusion of low-dose DEX during the night after surgery can significantly reduce the incidence of delirium, alleviate pain, and improve subjective sleep quality.

However, it is currently unclear whether choosing DEX during anesthesia has any impact on mortality and mental disorders in older patients undergoing non-cardiac surgery.

Therefore, we utilized prospective research data from 7 centers in China to explore the relationship between intraoperative use of DEX and postoperative 12-month mortality and mental disorders. Propensity score-matching (PSM) and Inverse probability of treatment weighting (IPTW) were conducted, and subgroup analyses were also applied.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years old, regardless of gender
2. Patients undergoing general anaesthesia (combined sedation or intravenous general anaesthesia)
3. ASA level 1-3
4. Patients undergoing elective non-cardiac surgery, non-neurosurgery

Exclusion Criteria:

1. More than 20% missing data for covariates;
2. Postoperative admission to the intensive care unit (ICU) or death during follow-up;
3. Preoperative history of severe sleep disorder and taking related medication;
4. Have a history of severe anxiety or depression prior to surgery and taking relevant medication;
5. Severe hearing, speech and cognitive impairments that preclude access to follow-up visits

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (≥ 65 years) who underwent elective major non-cardiac surgery were considered to be initially eligible. Non-cardiac surgery departments included otolaryngology surgery, urinary surgery, gynecology, gastrointestinal surgery, orthopedic surgery, thoracic surgery and hepato-pancreato-biliary surgery.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality rate | up to 12 month
  the 12-month all-cause mortality

SECONDARY OUTCOMES:
The incidence of postoperative delirium | During hospitalization (up to 1 month)
  the incidence of postoperative delirium (3D-CAM scale).Delirium was defined as acute, transient, fluctuating, and usually reversible disturbances in attention, cognition, or attention level. It was assessed every 12 hours by trained nurses using the confusion assessment method (CAM).
The incidence of postoperative anxiety | Anxiety within 7 days of surgery
  The GAD-7 is a seven-item questionnaire for screening on the presence of generalized anxiety disorder and assessing its severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-one. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe anxiety. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of anxiety. Higher scores mean more anxiety.
The incidence of postoperative depression | Depression within 7 days of surgery
  Primary outcomes were depression Patient Health Questionnaire 9 (PHQ-9).The PHQ-9 is a nine-item questionnaire for screening on the presence of depressive symptoms and monitoring depression severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-seven. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe level of depression. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of depression. The higher the score, the worse the situation. The total score ranges from 0 to 27, and higher scores indicate more depressive symptoms.
Postoperative sleep disorders | within 6 months after surgery
  The Hamilton Depression Scale (HAMD) sleep-related data and the Pittsburgh sleep quality index (PSQI) were used to evaluate the postoperative sleep abnormalities of the patients.
Surgical related complications | within 12 months after surgery
  Surgery-related complications include cardiovascular, respiratory, pulmonary, digestive, urinary, neurological, infection, pain, and bleeding from the surgery.
Postoperative quality of life evaluation | within 12 months after surgery
  Five-dimensional health scale EQ-5D, the five-dimensional health scale consists of 5 dimensions: mobility, self-care, activities of daily living, pain or discomfort, anxiety or depression. Each dimension contains three levels: no difficulty, some difficulty, and extreme difficulty. Through the conversion of effect size, the respondents can make choices at the five dimensions and three levels in the questionnaire, and calculate the score of the five-dimensional health scale index.

CONTACTS AND LOCATIONS:
Overall Officials: WEIDONG MI, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hao X, Zhang Z, Yang L, Guo Y, Cao F, Cao J, Liu Y, Lou J, Xu Z, Cui Y, Bai Y, Gu X, Wang D, Cui Q, Zhou Z, Shen H, Sun J, Mi W, Tong L. Association of Dexmedetomidine With Postoperative Depressive Symptoms in Older Surgical Patients: A Prospective Multicenter Study. CNS Neurosci Ther. 2025 May;31(5):e70407. doi: 10.1111/cns.70407. PMID 40387522